CLINICAL TRIAL: NCT03198780
Title: A Home-based Intervention to Promote Mindful Breathing Awareness Through Pursed-lip Breathing Training for COPD Patients
Brief Title: Mindful Breathing Awareness Through Pursed-Lip Breathing Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Mindful Breathing Intervention
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breathing Awareness (Experimental): In the clinic, once patients are proficient with the proposed tool, they will (1) independently don the pulse oximeter, (2) use the prototype to perform the mindful breathing intervention. The whole session will last no longer than 60 minutes with 30 minutes for the consent and demonstrations, two minutes to don the study devices, 15 minutes to practice mindful breathing, and two minutes to doff the study devices. The mindful breathing portion will be divided into three sessions. Each session will last three minutes and display a different presentation of Heart Rate Coherence biofeedback.
  At home, after completing the in-clinic study, five patients will take the mindful breathing tool home for a week to practice pursed-lip breathing at least five times. They will don the study devices, perform the intervention, and doff study devices.
  Interventions: Other: Breathing Awareness

INTERVENTIONS:
Other: Breathing Awareness — Participants will use a pulse-oximeter and biofeedback app to guide them through pursed-lip breathing training.

SUMMARY:
To establish the feasibility of a tool that monitors and motivates people with COPD to complete training in mindful pursed-lip breathing to enhance pulmonary rehabilitation at home.

DETAILED DESCRIPTION:
For this pilot study patients who meet the conventional criteria for pulmonary rehabilitation at their clinical appointments will be recruited and scheduled to return for the study. After completing the informed consent, patients will be taught how to don and doff the pulse oximeter, the source of the heart rate and oxygen signals. Patients will participate in a demonstration on how to perform the intervention. Recruitment will continue until five patients have completed the pilot in a clinic setting. If necessary, the prototype will be modified and testing resumed. Once the prototype system has met the criteria for success in the clinic, five of patients will be asked to use the prototype at the clinic and to take it home for a week and perform the intervention at least five times.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥40 years old
* have a diagnosis of GOLD stage II, III, or IV COPD documented by pulmonary function testing
* have clinically significant breathlessness (breathless when walking on the level or walking a mild hill)
* be a current or previous smoker with at least 10 pack-years of cigarette smoking
* be hospitalized for an exacerbation of COPD.

Exclusion Criteria:

* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move out of the state, are not living in the healthcare area.
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Participant assessment of device feasibility | up to 1 week
  Participants in both arms will complete a subjective questionnaire to elicit information about their experience and opinions about the intervention

SECONDARY OUTCOMES:
Device Use Assessed by Pulse Oximetry Data | up to 1 week
  The system will track data on each patient's breathing pattern to assess whether they are following the program

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kramer, Ph.D, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No